CLINICAL TRIAL: NCT06887673
Title: Exploring the Impact of Montelukast, SPM, and/or Almond/Almond Oil Supplementation on Lipid Mediator Biosynthesis in Colorectal, Sarcomas, Brain Tumors, Endometrial, and Ovarian Cancer: A Pilot Study
Brief Title: Lipid Mediators & Cancer: Montelukast, SPM, and Almonds
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY006089
Record Dates: First submitted 2025-02-25; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Sarcoma; Brain Tumors; Endometrial Cancer; Ovarian Cancer
Keywords: Montelukast; Almonds/Almond oil; Specialized pro-resolving mediators; Tumor-associated macrophages; Lipid mediators; Colorectal cancer; Inflammation
MeSH Terms: conditions — Colorectal Neoplasms; Sarcoma; Brain Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Inflammation | interventions — montelukast; Tablets

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Arm 1 (Control) (Other): ARM 1: Participants in this arm will receive no study treatment other than the standard of care management for their cancer.
  Interventions: Other: No Interventions
- Arm 2A: Sports Pro Resolve 4 g (Experimental): ARM 2A: Participants in this arm will receive 4 tabs (2 g) in the morning and 4 tabs (2 g) in the evening for 2 weeks before surgery.
  Interventions: Dietary Supplement: Sports Pro Resolve 4 g
- Arm 2B: Double Wood SPM 4 g (Experimental): ARM 2B: Participants in this arm will receive 4 tabs (2 g) in the morning and 4 tabs (2 g) in the evening for 2 weeks before surgery.
  Interventions: Dietary Supplement: Double Wood SPM 4 g
- Arm 3: California Sweet Almonds- 20 (Skin-on, Unsalted and Unprocessed) (Experimental): ARM 3: Participants in this arm will receive 20 skin-on, unsalted, unprocessed California Sweet Almonds, consumed as 10 almonds twice per day, for 2 weeks prior to surgery.
  Interventions: Dietary Supplement: 20 California Sweet Almonds
- Arm 4: Montelukast 10 mg (Experimental): ARM 4: Participants in this arm will receive Montelukast 10 mg orally daily for 2 weeks before surgery.
  Interventions: Drug: Montelukast 10 Mg Oral Tablet
- Arm 5: Montelukast 10 mg and SPM supplement 4 g (Experimental): ARM 5: Participants in this arm will receive a combination of Montelukast 10 mg daily and the determined SPM supplement 4 g daily, depending on which supplement produce the most SPMs in plasma.
  Interventions: Combination Product: Montelukast 10 Mg Oral Tablet and SPM 4 g
- Arm 6: Cold-Pressed Almond Oil 30 milliliter (Experimental): ARM 6; Participants in this arm will receive 30 milliliter of cold-pressed almond oil every morning with breakfast for 2 weeks before surgery
  Interventions: Dietary Supplement: Cold- Pressed Almond Oil 30 mL

INTERVENTIONS:
Other: No Interventions — No study treatment other than the standard of care management.
  Arms: Arm 1 (Control)
Dietary Supplement: Sports Pro Resolve 4 g — Sports Pro Resolve 4 tabs (2 g) twice daily
  Arms: Arm 2A: Sports Pro Resolve 4 g
Dietary Supplement: Double Wood SPM 4 g — Double Wood SPM 4 tabs (2 g) twice daily
  Arms: Arm 2B: Double Wood SPM 4 g
Dietary Supplement: 20 California Sweet Almonds — 10 California Sweet Almonds twice daily
  Arms: Arm 3: California Sweet Almonds- 20 (Skin-on, Unsalted and Unprocessed)
Drug: Montelukast 10 Mg Oral Tablet — Montelukast 10 Mg Oral Tablet daily
  Arms: Arm 4: Montelukast 10 mg
Combination Product: Montelukast 10 Mg Oral Tablet and SPM 4 g — Montelukast 10 Mg Oral Tablet and SPM 4 g
  Arms: Arm 5: Montelukast 10 mg and SPM supplement 4 g
Dietary Supplement: Cold- Pressed Almond Oil 30 mL — Cold- Pressed Almond Oil 30 mL every morning
  Arms: Arm 6: Cold-Pressed Almond Oil 30 milliliter

SUMMARY:
The purpose of this study is to create a prospective investigation to examine the effects of montelukast, almonds/almond oil, and specialized pro-resolving mediators (SPMs) on lipid profiles and tumor-associated macrophages (TAMs) in cancer patients (colorectal cancer, sarcoma, brain tumors, endometrial cancer, and ovarian cancer). The focus will be on assessing changes in lipid mediator concentrations, TAM reprogramming, and immune cell function in treated versus untreated patients. It is hypothesized that montelukast will reduce the pro-inflammatory effects of leukotriene B4 (LTB4), while SPMs and almonds/almond oil will shift the balance toward pro-resolving mediators, enhancing anti-inflammatory and immune-stimulatory responses and reprogramming TAMs.

DETAILED DESCRIPTION:
This prospective study investigates the effects of montelukast, almonds/almond oil, and specialized pro-resolving mediators (SPMs) on lipid profiles and tumor-associated macrophages (TAMs) in patients with colorectal cancer (CRC), sarcoma, brain tumors (BT), endometrial cancer (EC), and ovarian cancer (OvCa). Patients receiving these treatments will be compared to untreated controls, with tissue samples collected post-surgery for analysis. A cohort of patients who have undergone tumor resection will be included for the assessment of lipid mediator concentrations (approximately 65 arachidonic acid pathway lipids) and TAM reprogramming, with an emphasis on comparing treated and untreated groups. The study will also examine peripheral blood mononuclear cells (PBMCs) and plasma concentrations of lipid mediators before and after treatment, focusing on changes in PBMC function and phenotype. It is hypothesized that montelukast, an LTB4/ cysteinyl leukotriene receptor 1 (CYSLTR1) inhibitor, will reduce the pro-inflammatory effects of LTB4 in cancer tissues. Furthermore, it is anticipated that SPMs and almonds/almond oil will shift the lipid mediator balance toward pro-resolving mediators, enhancing anti-inflammatory responses, stimulating immune function, and reprogramming TAMs.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed individuals with stages I-IV colorectal or ovarian cancer, grade 1 and 2 endometrial cancer, as well as those with brain tumors or sarcoma.
2. Participants scheduled for surgical intervention at least two (2) weeks from the day of enrollment.
3. Patients must be able to understand and willing to sign a written informed consent document for both this study and the University of South Florida (USF)/ Tampa General Hospital (TGH) Biorepository study (STUDY000356).
4. Age 18 or older.

Exclusion Criteria:

1. Inability to give consent due to a mental condition that makes the participant unable to understand the study's nature, scope, and possible consequences.
2. Participants who are unlikely to adhere to the protocol as determined by the study investigator.
3. Allergy to fish, seafood, aspirin, NSAIDs, montelukast, or nuts
4. Participants with a history of asthma or chronic obstructive pulmonary disease (COPD).
5. Patients with a history of phenylketonuria (PKU).
6. Participants with a history of a psychiatric illness (e.g., major depression, anxiety disorder, bipolar disorder, obsessive-compulsive disorder, etc.).
7. Surgical intervention scheduled more than eight (8) weeks from the initial enrollment day.
8. No evidence of a discrete mass on endoscopy or radiologic imaging
9. Concomitant existence of other malignancies
10. Uncontrolled hypertension or diabetes mellitus
11. Chronic Liver Disease or cirrhosis
12. Liver function impairment or persisting elevations (confirmed by retest) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or direct bilirubin greater than 2x the upper limit of the normal range (ULN)
13. Bleeding conditions such as disorders of platelet function, idiopathic thrombocytopenia purpura (ITP), thrombotic thrombocytopenic purpura (TTP), hemophilia or any clotting factor deficiency, von Willebrand disease or Glanzmann disease among other
14. Use of antiplatelet or anticoagulant medications, including aspirin, clopidogrel, warfarin, direct oral anticoagulants (DOACs), and heparin, among others
15. Persistent significant or severe infection, either acute or chronic
16. Participants with significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia (confirmed by retest):

    1. Hematocrit < 35% and/or
    2. Absolute white blood cell count < 3000 cells/mm3 (μL) and/or
    3. Platelet count < 150 000 cells/mm3 (μL) and/or
    4. Absolute neutrophil ≤ 1500 cells/mm3 (μL)
17. Chronic use of immunosuppressive medications
18. History of organ transplantation
19. Emergency surgery
20. Pregnant or breast-feeding women or those who plan to become pregnant during the study.
21. Women of childbearing potential who are not protected by effective contraceptive methods of birth control and/or are unwilling or unable to be tested for pregnancy.
22. Prisoners
23. Participants who have received treatment with leukotriene inhibitors, taken omega-3 supplements, or eaten almonds within the last 4 weeks.
24. Prior use of any investigational drug in the preceding six (6) months
25. Participants who, after being enrolled in this study and assigned a particular study treatment, consume products involved in other study cohorts other than what they were assigned (i.e. if a patient is assigned to take SPMs as their study treatment but during the course of the study also is consuming daily almonds)
26. Participants who are unable to swallow oral medication or chew almonds.
27. Participants who have already started neoadjuvant therapies for their cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quantity of lipid mediators in a tumor specimen after 2 weeks of study treatment. | Day 14 of treatment
  Quantitation will be assessed using liquid chromatography tandem mass spectrometry (LC-MS/MS). The absolute quantity of these lipid mediators will be compared to the absolute quantity in the corresponding normal tissue. In preliminary studies, the investigators have used LC-MS/MS to measure ~65 different lipid mediators of the arachidonic acid pathway in colorectal cancer. Interestingly, the investigators found high proportions of pro-inflammation mediators and depressed levels of pro-resolution-of-inflammation mediators in cancer tissue compared with the non-affected tissue of the same patients. Possible study treatments include: specialized pro-resolving mediators vs Montelukast vs almonds/almond oil vs combination).
Quantity of lipid mediators in a non-cancerous (i.e. normal) tissue from the resected surgical specimen after 2 weeks of study treatment. | Day 14 of treatment
  Quantitation will be assessed using liquid chromatography tandem mass spectrometry (LC-MS/MS). The absolute quantity of these lipid mediators will be compared to the absolute quantity in the corresponding cancer tissue. This change in quantity will enable us to make deductions about the influence of the corresponding study treatment on the tumor and its environment. For example, does the treatment in question make the tumor environment less inflamed/promote healing and therefore make the cancer more susceptible to treatment? Possible study treatments include: specialized pro-resolving mediators vs Montelukast vs almonds/almond oil vs combination).

SECONDARY OUTCOMES:
Quantity of tumor microenvironment subpopulations in a tumor specimen versus corresponding normal tissue after 2 weeks of study treatment. | Day 14 of treatment
  Tumor microenvironment subpopulations are defined as the various components of the immune system in the tissue surrounding a cancer, i.e.: cluster of differentiation 4 (CD4) T cells, cluster of differentiation 8 (CD8) T cells, B cells, natural killer (NK) cells, macrophages, etc. Quantitation will be assessed using n-counter analysis.
Distribution of tumor-associated macrophage (TAM) phenotype in tumor specimens versus corresponding normal tissue after 2 weeks of study treatment. | Day 14 of treatment
  There are two main TAM phenotypes: M1 and M2. M1 are the classically activated, anti-tumor macrophages, and M2 are the "bad", pro-inflammation/neoplastic macrophages. Change in distribution will be assessed using multiparameter flow cytometry. M1 versus M2 phenotypes will be identified by utilizing macrophage-specific biomarkers.
Functionality of tumor-associated macrophages in tumor specimens versus corresponding normal tissue after 2 weeks of study treatment. | Day 14 of treatment
  Change in functionality will be determined using efferocytosis assays.
Change in quantity of lipids in peripheral blood from day 0 to day 14 of study treatment. | Day 0 and Day 14
  Quantitation will be assessed using liquid chromatography tandem mass spectrometry (LC-MS/MS). This assessment will enable us to correlate peripheral blood levels of lipid mediators with tissue penetrance. For example, the investigators may find that a study treatment has a significant impact on the lipid mediator profile of the blood but that same impact is not seen in the corresponding tissue of that patient; therefore, there deductions can be made about tissue penetrance capability.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Marcet, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad S, Sung B, Aggarwal BB. Age-associated chronic diseases require age-old medicine: role of chronic inflammation. Prev Med. 2012 May;54 Suppl(Suppl):S29-37. doi: 10.1016/j.ypmed.2011.11.011. Epub 2011 Dec 9. PMID 22178471
- [Background] Serhan CN. Discovery of specialized pro-resolving mediators marks the dawn of resolution physiology and pharmacology. Mol Aspects Med. 2017 Dec;58:1-11. doi: 10.1016/j.mam.2017.03.001. Epub 2017 Mar 3. PMID 28263773
- [Background] Song M, Zhang X, Meyerhardt JA, Giovannucci EL, Ogino S, Fuchs CS, Chan AT. Marine omega-3 polyunsaturated fatty acid intake and survival after colorectal cancer diagnosis. Gut. 2017 Oct;66(10):1790-1796. doi: 10.1136/gutjnl-2016-311990. Epub 2016 Jul 19. PMID 27436272
- [Background] Daniel CR, McCullough ML, Patel RC, Jacobs EJ, Flanders WD, Thun MJ, Calle EE. Dietary intake of omega-6 and omega-3 fatty acids and risk of colorectal cancer in a prospective cohort of U.S. men and women. Cancer Epidemiol Biomarkers Prev. 2009 Feb;18(2):516-25. doi: 10.1158/1055-9965.EPI-08-0750. Epub 2009 Feb 3. PMID 19190143
- [Background] Shin A, Cho S, Sandin S, Lof M, Oh MY, Weiderpass E. Omega-3 and -6 Fatty Acid Intake and Colorectal Cancer Risk in Swedish Women's Lifestyle and Health Cohort. Cancer Res Treat. 2020 Jul;52(3):848-854. doi: 10.4143/crt.2019.550. Epub 2020 Mar 6. PMID 32138465
- [Background] Schloss I, Kidd MS, Tichelaar HY, Young GO, O'Keefe SJ. Dietary factors associated with a low risk of colon cancer in coloured west coast fishermen. S Afr Med J. 1997 Feb;87(2):152-8. PMID 9107220
- [Background] Petrik MB, McEntee MF, Chiu CH, Whelan J. Antagonism of arachidonic acid is linked to the antitumorigenic effect of dietary eicosapentaenoic acid in Apc(Min/+) mice. J Nutr. 2000 May;130(5):1153-8. doi: 10.1093/jn/130.5.1153. PMID 10801912
- [Background] Fini L, Piazzi G, Ceccarelli C, Daoud Y, Belluzzi A, Munarini A, Graziani G, Fogliano V, Selgrad M, Garcia M, Gasbarrini A, Genta RM, Boland CR, Ricciardiello L. Highly purified eicosapentaenoic acid as free fatty acids strongly suppresses polyps in Apc(Min/+) mice. Clin Cancer Res. 2010 Dec 1;16(23):5703-11. doi: 10.1158/1078-0432.CCR-10-1990. Epub 2010 Oct 28. PMID 21030497
- [Background] Nowak J, Weylandt KH, Habbel P, Wang J, Dignass A, Glickman JN, Kang JX. Colitis-associated colon tumorigenesis is suppressed in transgenic mice rich in endogenous n-3 fatty acids. Carcinogenesis. 2007 Sep;28(9):1991-5. doi: 10.1093/carcin/bgm166. Epub 2007 Jul 18. PMID 17634405
- [Background] West NJ, Clark SK, Phillips RK, Hutchinson JM, Leicester RJ, Belluzzi A, Hull MA. Eicosapentaenoic acid reduces rectal polyp number and size in familial adenomatous polyposis. Gut. 2010 Jul;59(7):918-25. doi: 10.1136/gut.2009.200642. Epub 2010 Mar 26. PMID 20348368
- [Background] Liang B, Wang S, Ye YJ, Yang XD, Wang YL, Qu J, Xie QW, Yin MJ. Impact of postoperative omega-3 fatty acid-supplemented parenteral nutrition on clinical outcomes and immunomodulations in colorectal cancer patients. World J Gastroenterol. 2008 Apr 21;14(15):2434-9. doi: 10.3748/wjg.14.2434. PMID 18416476
- [Background] Sorensen LS, Thorlacius-Ussing O, Rasmussen HH, Lundbye-Christensen S, Calder PC, Lindorff-Larsen K, Schmidt EB. Effects of perioperative supplementation with omega-3 fatty acids on leukotriene B(4) and leukotriene B(5) production by stimulated neutrophils in patients with colorectal cancer: a randomized, placebo-controlled intervention trial. Nutrients. 2014 Sep 29;6(10):4043-57. doi: 10.3390/nu6104043. PMID 25268838
- [Background] Manda K, Kriesen S, Hildebrandt G, Fietkau R, Klautke G. Omega-3 fatty acid supplementation in cancer therapy : does eicosapentanoic acid influence the radiosensitivity of tumor cells? Strahlenther Onkol. 2011 Feb;187(2):127-34. doi: 10.1007/s00066-010-2166-6. Epub 2011 Jan 18. PMID 21267532
- [Background] West L, Yin Y, Pierce SR, Fang Z, Fan Y, Sun W, Tucker K, Staley A, Zhou C, Bae-Jump V. Docosahexaenoic acid (DHA), an omega-3 fatty acid, inhibits tumor growth and metastatic potential of ovarian cancer. Am J Cancer Res. 2020 Dec 1;10(12):4450-4463. eCollection 2020. PMID 33415010
- [Background] Kuznetsova L, Chen J, Sun L, Wu X, Pepe A, Veith JM, Pera P, Bernacki RJ, Ojima I. Syntheses and evaluation of novel fatty acid-second-generation taxoid conjugates as promising anticancer agents. Bioorg Med Chem Lett. 2006 Feb 15;16(4):974-7. doi: 10.1016/j.bmcl.2005.10.089. Epub 2005 Nov 18. PMID 16298526
- [Background] Wang YC, Wu YN, Wang SL, Lin QH, He MF, Liu QL, Wang JH. Docosahexaenoic Acid Modulates Invasion and Metastasis of Human Ovarian Cancer via Multiple Molecular Pathways. Int J Gynecol Cancer. 2016 Jul;26(6):994-1003. doi: 10.1097/IGC.0000000000000746. PMID 27258728
- [Background] Wen Z, Liu H, Li M, Li B, Gao W, Shao Q, Fan B, Zhao F, Wang Q, Xie Q, Yang Y, Yu J, Qu X. Increased metabolites of 5-lipoxygenase from hypoxic ovarian cancer cells promote tumor-associated macrophage infiltration. Oncogene. 2015 Mar 5;34(10):1241-52. doi: 10.1038/onc.2014.85. Epub 2014 Mar 24. PMID 24662827
- [Background] Wang Y, Liu K, Long T, Long J, Li Y, Li J, Cheng L. Dietary fish and omega-3 polyunsaturated fatty acids intake and cancer survival: A systematic review and meta-analysis. Crit Rev Food Sci Nutr. 2023;63(23):6235-6251. doi: 10.1080/10408398.2022.2029826. Epub 2022 Jan 24. PMID 35068276
- [Background] Jang HY, Kim IW, Oh JM. Cysteinyl Leukotriene Receptor Antagonists Associated With a Decreased Incidence of Cancer: A Retrospective Cohort Study. Front Oncol. 2022 Apr 7;12:858855. doi: 10.3389/fonc.2022.858855. eCollection 2022. PMID 35463337
- [Background] Higurashi T, Ashikari K, Tamura S, Saigusa Y, Takatsu T, Misawa N, Yoshihara T, Matsuura T, Fuyuki A, Ohkubo H, Kessoku T, Hosono K, Yoneda M, Nakajima A. Leukotriene Receptor Antagonist Therapy for the Chemoprevention of Human Rectal Aberrant Crypt Foci: Nonrandomized, Open-Label, Controlled Trial. Cancer Prev Res (Phila). 2022 Oct 4;15(10):661-668. doi: 10.1158/1940-6207.CAPR-22-0049. PMID 36083855
- [Background] Lien EL. Toxicology and safety of DHA. Prostaglandins Leukot Essent Fatty Acids. 2009 Aug-Sep;81(2-3):125-32. doi: 10.1016/j.plefa.2009.05.004. Epub 2009 Jun 6. PMID 19501496
- [Background] Villani AM, Crotty M, Cleland LG, James MJ, Fraser RJ, Cobiac L, Miller MD. Fish oil administration in older adults: is there potential for adverse events? A systematic review of the literature. BMC Geriatr. 2013 May 1;13:41. doi: 10.1186/1471-2318-13-41. PMID 23634646
- [Background] Souza PR, Marques RM, Gomez EA, Colas RA, De Matteis R, Zak A, Patel M, Collier DJ, Dalli J. Enriched Marine Oil Supplements Increase Peripheral Blood Specialized Pro-Resolving Mediators Concentrations and Reprogram Host Immune Responses: A Randomized Double-Blind Placebo-Controlled Study. Circ Res. 2020 Jan 3;126(1):75-90. doi: 10.1161/CIRCRESAHA.119.315506. Epub 2019 Dec 12. PMID 31829100
- [Background] FDA. FDA requires stronger warning about risk of neuropsychiatric events associated with asthma and allergy drug montelukast. . Published March 4, 2020. Accessed February 18, 2023. https://www.fda.gov/news-events/press-announcements/fda-requires-stronger-warning-about-risk-neuropsychiatric-events-associated-asthma-and-allergy
- [Background] Aldea Perona A, Garcia-Saiz M, Sanz Alvarez E. Psychiatric Disorders and Montelukast in Children: A Disproportionality Analysis of the VigiBase((R)). Drug Saf. 2016 Jan;39(1):69-78. doi: 10.1007/s40264-015-0360-2. PMID 26620206
- [Background] Benard B, Bastien V, Vinet B, Yang R, Krajinovic M, Ducharme FM. Neuropsychiatric adverse drug reactions in children initiated on montelukast in real-life practice. Eur Respir J. 2017 Aug 17;50(2):1700148. doi: 10.1183/13993003.00148-2017. Print 2017 Aug. PMID 28818882
- [Background] Ali MM, O'Brien CE, Cleves MA, Martin BC. Exploring the possible association between montelukast and neuropsychiatric events among children with asthma: a matched nested case-control study. Pharmacoepidemiol Drug Saf. 2015 Apr;24(4):435-45. doi: 10.1002/pds.3758. Epub 2015 Feb 12. PMID 25683909
- [Background] Sansing-Foster V, Haug N, Mosholder A, Cocoros NM, Bradley M, Ma Y, Pennap D, Dee EC, Toh S, Pestine E, Petrone AB, Kim I, Lyons JG, Eworuke E. Risk of Psychiatric Adverse Events Among Montelukast Users. J Allergy Clin Immunol Pract. 2021 Jan;9(1):385-393.e12. doi: 10.1016/j.jaip.2020.07.052. Epub 2020 Aug 11. PMID 32795564
- [Background] Knapp HR, Reilly IA, Alessandrini P, FitzGerald GA. In vivo indexes of platelet and vascular function during fish-oil administration in patients with atherosclerosis. N Engl J Med. 1986 Apr 10;314(15):937-42. doi: 10.1056/NEJM198604103141501. PMID 3007982
- [Background] Abdelhamid AS, Brown TJ, Brainard JS, Biswas P, Thorpe GC, Moore HJ, Deane KH, Summerbell CD, Worthington HV, Song F, Hooper L. Omega-3 fatty acids for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Feb 29;3(3):CD003177. doi: 10.1002/14651858.CD003177.pub5. PMID 32114706
- [Background] Akintoye E, Sethi P, Harris WS, Thompson PA, Marchioli R, Tavazzi L, Latini R, Pretorius M, Brown NJ, Libby P, Mozaffarian D. Fish Oil and Perioperative Bleeding. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004584. doi: 10.1161/CIRCOUTCOMES.118.004584. PMID 30571332
- [Background] Mozaffarian D, Rimm EB. Fish intake, contaminants, and human health: evaluating the risks and the benefits. JAMA. 2006 Oct 18;296(15):1885-99. doi: 10.1001/jama.296.15.1885. PMID 17047219
- [Background] Nicholls SJ, Lincoff AM, Garcia M, Bash D, Ballantyne CM, Barter PJ, Davidson MH, Kastelein JJP, Koenig W, McGuire DK, Mozaffarian D, Ridker PM, Ray KK, Katona BG, Himmelmann A, Loss LE, Rensfeldt M, Lundstrom T, Agrawal R, Menon V, Wolski K, Nissen SE. Effect of High-Dose Omega-3 Fatty Acids vs Corn Oil on Major Adverse Cardiovascular Events in Patients at High Cardiovascular Risk: The STRENGTH Randomized Clinical Trial. JAMA. 2020 Dec 8;324(22):2268-2280. doi: 10.1001/jama.2020.22258. PMID 33190147
- [Background] Nielsen CK, Ohd JF, Wikstrom K, Massoumi R, Paruchuri S, Juhas M, Sjolander A. The leukotriene receptor CysLT1 and 5-lipoxygenase are upregulated in colon cancer. Adv Exp Med Biol. 2003;525:201-4. doi: 10.1007/978-1-4419-9194-2_43. No abstract available. PMID 12751768
- [Background] Burke L, Butler CT, Murphy A, Moran B, Gallagher WM, O'Sullivan J, Kennedy BN. Evaluation of Cysteinyl Leukotriene Signaling as a Therapeutic Target for Colorectal Cancer. Front Cell Dev Biol. 2016 Sep 21;4:103. doi: 10.3389/fcell.2016.00103. eCollection 2016. PMID 27709113
- [Background] Sulciner ML, Serhan CN, Gilligan MM, Mudge DK, Chang J, Gartung A, Lehner KA, Bielenberg DR, Schmidt B, Dalli J, Greene ER, Gus-Brautbar Y, Piwowarski J, Mammoto T, Zurakowski D, Perretti M, Sukhatme VP, Kaipainen A, Kieran MW, Huang S, Panigrahy D. Resolvins suppress tumor growth and enhance cancer therapy. J Exp Med. 2018 Jan 2;215(1):115-140. doi: 10.1084/jem.20170681. Epub 2017 Nov 30. PMID 29191914
- [Background] Ahmad Z. The uses and properties of almond oil. Complement Ther Clin Pract. 2010 Feb;16(1):10-2. doi: 10.1016/j.ctcp.2009.06.015. Epub 2009 Jul 15. PMID 20129403
- [Background] Mericli F, Becer E, Kabadayi H, Hanoglu A, Yigit Hanoglu D, Ozkum Yavuz D, Ozek T, Vatansever S. Fatty acid composition and anticancer activity in colon carcinoma cell lines of Prunus dulcis seed oil. Pharm Biol. 2017 Dec;55(1):1239-1248. doi: 10.1080/13880209.2017.1296003. PMID 28262033
- [Background] Hollis J, Mattes R. Effect of chronic consumption of almonds on body weight in healthy humans. Br J Nutr. 2007 Sep;98(3):651-6. doi: 10.1017/S0007114507734608. Epub 2007 Apr 20. PMID 17445351
- [Background] Ali ZK, Sahib HB. Antiangiogenic Activity of Sweet Almond (Prunus dulcis) Oil Alone and in Combination with Aspirin in both in vivo and in vitro Assays. Asian Pac J Cancer Prev. 2022 Apr 1;23(4):1405-1413. doi: 10.31557/APJCP.2022.23.4.1405. PMID 35485703
- [Background] Hyson DA, Schneeman BO, Davis PA. Almonds and almond oil have similar effects on plasma lipids and LDL oxidation in healthy men and women. J Nutr. 2002 Apr;132(4):703-7. doi: 10.1093/jn/132.4.703. PMID 11925464
- [Background] Fraser GE, Sabate J, Beeson WL, Strahan TM. A possible protective effect of nut consumption on risk of coronary heart disease. The Adventist Health Study. Arch Intern Med. 1992 Jul;152(7):1416-24. PMID 1627021
- [Background] Dreher ML. A Comprehensive Review of Almond Clinical Trials on Weight Measures, Metabolic Health Biomarkers and Outcomes, and the Gut Microbiota. Nutrients. 2021 Jun 8;13(6):1968. doi: 10.3390/nu13061968. PMID 34201139
- [Background] Aune D, Keum N, Giovannucci E, Fadnes LT, Boffetta P, Greenwood DC, Tonstad S, Vatten LJ, Riboli E, Norat T. Nut consumption and risk of cardiovascular disease, total cancer, all-cause and cause-specific mortality: a systematic review and dose-response meta-analysis of prospective studies. BMC Med. 2016 Dec 5;14(1):207. doi: 10.1186/s12916-016-0730-3. PMID 27916000